CLINICAL TRIAL: NCT07323524
Title: Sodium-Glucose Co-Transporter-2 Inhibitors in Lupus Nephritis
Brief Title: Dapagliflozin in Active Lupus Nephritis
Acronym: Dapa-Active LN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen H. Costenbader, Associate Physician, Rheumatologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P003238
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis (LN)
Keywords: dapagliflozin; SGLT2 inhibitor; safety; feasibility; pilot trial
MeSH Terms: conditions — Lupus Nephritis | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: Pilot and feasibility, concealed allocation, blinded randomized controlled trial of dapagliflozin 10 mg/day or matched placebo in a 2:1 allocation ratio (22 subjects active arm: 11 subjects placebo arm), in addition to standard-of-care treatment, for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg daily (Active Comparator): Subjects will receive masked dapagliflozin 10 mg daily for 12 weeks
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy
- Matching placebo pill daily (Placebo Comparator): Subjects will receive a matching placebo pill to take daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Pilot and feasibility of adding dapagliflozin to standard medical therapy in active lupus nephritis (LN)
  Arms: Dapagliflozin 10 mg daily
Drug: Placebo — Matching placebo daily with standard of care
  Arms: Matching placebo pill daily

SUMMARY:
Lupus nephritis is a chronic and life-threatening autoimmune cause of kidney disease that predominately impacts young people and can lead to kidney failure. Sodium-glucose co-transporter-2 inhibitors, including dapagliflozin, are known to improve outcomes for people with other causes of chronic kidney disease. This pilot and feasibility randomized clinical trial will test the use of dapagliflozin versus placebo in addition to standard of care treatment for patients with early and active lupus nephritis, a group who has not been included in past trials.

DETAILED DESCRIPTION:
This is a pilot and feasibility randomized, double-blind, placebo-controlled trial involving patients with active lupus nephritis. It will be a concealed allocation, blinded randomized controlled trial of dapagliflozin 10 mg/day or matched placebo in a 2:1 allocation ratio (22 subjects active arm: 11 subjects placebo arm), in addition to standard-of-care treatment, for 12 weeks. After informed consent, 33 eligible subjects will be randomized 2:1 to oral dapagliflozin 10 mg/day or identical oral placebo/day for 12 weeks. Study visits will occur at screening (Visit -1), baseline (Visit 0) and weeks 4 (Visit 1), 8 (Visit 2) and 12 (Visit 3). Observational data including laboratory test results obtained in routine clinical care will be collected through 12 months of follow-up.

The primary outcomes are:

1. the overall proportion of identified as potentially eligible/pre-screened patients who enroll in the trial;
2. feasibility and completeness of data collection procedures;
3. changes in urine protein-to-creatinine ratio (UPCR) and precision of these estimates from baseline to week 12 in each group; and
4. rates and proportions of serious adverse events and of adverse events of interest, including genitourinary infections and volume depletion.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-70 years, fulfilling 2012 SLICC or 2019 ACR/EULAR criteria for SLE, with biopsy-proven class III, IV and/or V LN

  * Active (new or relapsing) LN within the prior six months, with at least one of the following:

    * Kidney biopsy with activity index >2 and/or
    * Active urinary sediment (>5 RBCs, >5 WBCs, or cellular casts)
  * Receiving standard-of-care immunosuppression regimen for active LN, including mycophenolate, cyclophosphamide, belimumab, azathioprine, a calcineurin inhibitor, and/or B cell depleting therapies
  * Recent or ongoing glucocorticoids use for active LN within the past 6 months
  * Receiving standard-of-care antimalarial therapy and RAAS blockade, unless contraindicated
  * Estimated ≥0.5 g/g 24 hr proteinuria or ≥0.3 mg/g 24 hr microalbuminuria at enrollment (on first morning urine)
  * Ability to given informed consent

Exclusion Criteria:

* GFR < 25 ml/min/1.73m2

  * Acute kidney injury at study enrollment (>50 percent rise in creatinine within 90 days)
  * Type I diabetes, underweight (BMI <18.5), active malignancy, active infection, or recurrent genitourinary infections
  * For females: pregnancy, or desiring of pregnancy and not using contraception, or unable to use contraception
  * Current use of >1mg/kg/day prednisone equivalent
  * Current or prior use of SGLT2 inhibitors or GLP-1 receptor agonists

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible enrolled | 3 years
  The overall proportion of identified as potentially eligible/pre-screened patients who enroll in the trial

SECONDARY OUTCOMES:
Feasibility of data collection | 3 years
  We will assess the percent of missing data elements overall at pilot trial completion.

OTHER OUTCOMES:
Change in urine protein-to-creatinine ratio | 12 weeks per subject
  Change in urine protein-to-creatinine ratio (UPCR) from baseline to week 12 in each group
Adverse outcomes | 3 years
  Rates and proportions of serious adverse events and of adverse events of interest, including genitourinary infections and volume depletion

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts